CLINICAL TRIAL: NCT06382623
Title: Comparing the Effectiveness of Peritendinous Steroid Injection Under Ultrasound Guidance With Percutaneous A1 Pulley Release in Trigger Finger Treatment
Brief Title: Efficacies of Different Managements in Patients With Trigger Finger
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, principal investigator, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 43
Record Dates: First submitted 2024-04-08; First posted 2024-04-24 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The peritendinous steroid group: A 1 ml mixture of corticosteroid (2 mg + 5 mg/ml betamethasone) and 1 ml of local anesthetic agent (20 ml 2% prilocaine) was injected peritendinously between the A1 pulley and the flexor tendon sheath at the metacarpophalangeal joint level under ultrasound guidance.
  Interventions: Other: The peritendinous Betamethasone group
- The percutaneous A1 pulley release group: In the A1 pulley release group, 1 ml of local anesthetic agent (20 ml 2% prilocaine) was injected into the pulley-associated subcutaneous tissue using a 27 G needle under ultrasound guidance. The metacarpophalangeal joint was brought into slight hyperextension. Subsequently, a 20 G 0.9x38mm needle, modified by bending approximately 40-45 degrees from the proximal 1/3 of the needle with the aid of a cap, was used. The needle was advanced in-plane from distal to proximal along the midline, with simultaneous movement towards the palmar surface, aiming to cut or loosen the pulley between the tendon and A1 pulley. The loosening procedure was repeated from the distal to proximal aspect of the pulley until the sensation of resistance at the needle tip disappeared.
  Interventions: Procedure: The percutaneous A1 pulley release

INTERVENTIONS:
Procedure: The percutaneous A1 pulley release — Ultrasound-guided percutaneous pulley release is a procedure aimed at loosening the pulley using various cutting instruments or hypodermic needles under ultrasound guidance.
  Groups: The percutaneous A1 pulley release group
Other: The peritendinous Betamethasone group — USG-guided injection of corticosteroid between the A1 pulley and the flexor tendon sheath.
  Groups: The peritendinous steroid group

SUMMARY:
The aim of the study is to compare the effectiveness of peritendinous steroid injection under ultrasound guidance and percutaneous A1 pulley release procedures in terms of disease stage, pain, and severity of locking in patients with trigger finger.

DETAILED DESCRIPTION:
This study was designed as a randomized, controlled, prospective study. Patients who had been experiencing trigger finger symptoms for at least one month and who presented to the Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, affiliated with the Health Sciences University Faculty of Medicine

Patients were randomly divided into two groups: the peritendinous steroid group (n=15) and the percutaneous pulley release group (n=15). In the first group, under ultrasound guidance, a mixture of 1 ml corticosteroid (2 mg+5 mg/ml betamethasone) and 1 ml local anesthetic (20 ml 2% prilocaine) was injected peritendinously between the A1 pulley and the flexor tendon sheath. In the second group, a percutaneous A1 pulley release procedure was performed under ultrasound guidance using a 20 G needle, followed by peritendinous injection of the same mixture of corticosteroid and local anesthetic.

Patients were evaluated four times: before treatment, at 1 week, 1 month, and 3 months after treatment. Modified Quinnel classification, VAS (Visual Analog Scale), and severity of locking scales were used as outcome measures in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age
* Having had trigger finger complaints for more than 1 month
* Not having received any injections for trigger finger diagnosis within the last 1 month
* Signing the informed consent form indicating willingness to participate in the study

Exclusion Criteria:

* Refusing to participate in the study
* Presence of partial or complete tendon rupture in the relevant tendon of the finger to be treated
* Presence of wounds and infection in the area where the procedure will be performed
* Pregnancy status
* History of allergy to the injected medications (local anesthetic, steroid)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: older 18 ages
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Stage of the disease | first week, first mount, third month
  Modified Quinnel classification Stage 1: Normal movement, no pain.
  * Stage 2: Normal movement, occasional pain.
  * Stage 3: Irregular movement (catching without crepitus or locking).
  * Stage 4: Locking present, actively correctable.
  * Stage 5: Locking present, passively correctable.

SECONDARY OUTCOMES:
Pain intensity | first week, first month, third month
  The pain associated with movement in the relevant finger was evaluated using the Visual Analog Scale (VAS). Patients were explained that "0" represented no pain at all, "10" represented the most severe pain they had ever experienced in their life, and "5" represented moderate pain. They were asked to indicate a number between 0 and 10 that corresponded to the intensity of pain they were feeling.
severity of triggering | first week, first month, third month
  The severity of catching in patients was assessed using a Numeric Rating Scale (NRS) ranging from 0 to 10. Patients were explained that "0" represents no catching at all, while "10" represents catching requiring passive correction of the finger. They were asked to mark a number between 0 and 10 corresponding to the severity of catching they experienced.

CONTACTS AND LOCATIONS:
Overall Officials: zeliha gizem mac, MD, Principal Investigator — university of health sciences, Department of PM&R
Locations (1):
- Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No